CLINICAL TRIAL: NCT02557126
Title: A Placebo-controlled, Randomized, Double-blind, Multicenter Phase 2 Study to Assess the Efficacy and Safety of URC102 in Gout Patients
Brief Title: Study of URC102 to Assess the Safety and Efficacy in Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URC103KR
Record Dates: First submitted 2015-09-16; First posted 2015-09-23 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — URC102

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- URC102 (Experimental): URC102
  Interventions: Drug: URC102
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: URC102
  Arms: URC102
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety, Pharmacokinetics/Pharmacodynamics and Urate Lowering Effect of URC102 in gout patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gout

Exclusion Criteria:

* Participated in other clinical study within 12 weeks prior to enrollment, and received an investigational product (including placebo)

Ages: 20 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Trend of serum uric acid reduction rate (%) | 2 weeks
Trend of serum uric acid levels (mg/dL) | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- JW Pharmaceutical, Seoul, Seocho-dong, South Korea